CLINICAL TRIAL: NCT05062018
Title: Vitamin D3 - Omega3 - Home Exercise - HeALTHy Aging and Longevity Cohort
Acronym: DO-HEALTH-C
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Heike Bischoff-Ferrari (Other)
Responsible Party: Sponsor-Investigator, Heike Bischoff-Ferrari, Prof. Dr. med. DrPH, University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: 2019-00134
Record Dates: First submitted 2021-09-20; First posted 2021-09-30 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Healthy Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The DO-HEALTH trial will be extended into the cohort including the collection on life style factors such as diet, quality of life and physical activity, as well as health-related data on co-morbid conditions as well as a standardized assessment of multiple organ functions, physical, cognitive and mental function using surveys and standardized health assessments.

DETAILED DESCRIPTION:
The DO-HEALTH cohort will be a continuation of the trial without intervention and will elucidate longterm determinants of healthy, active and independent aging in European community-dwelling older adults. The main emphasize of the cohort will be to determine the risk factors, to quantify the incidence and to describe the trajectories of incident frailty, impaired mobility, loss of independence and age related morbidity (e.g. heart arrhythmia, type 2 diabetes, falls, fractures).

Additionally, the cohort will continue to investigate the primary endpoints of the original trial like the risk and incidence of injurious falls (bone); functional decline (muscle); high blood pressure (cardiovascular); cognitive decline (brain); and the rate of any infection (immunity). Moreover, the cohort will include and extend key secondary and exploratory endpoints of the original trial such as incidence and prevalence of anemia, sarcopenia, cardiovascular diseases, type 2 diabetes and cancer.

ELIGIBILITY:
Inclusion Criteria:

* Former participation in the DO-HEALTH clinical trial study

Exclusion Criteria:

* Inability or unwillingness to give written informed consent
* Medical condition that would make the results of the tests/assessments unreliable and/or would put too much burden to the participant, and/or leads to safety concerns.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The DO-HEALTH Cohort includes the population of the former DO-HEALTH clinical trial (NCT01745263)
Sampling Method: Non-Probability Sample
Enrollment: 534 (Estimated)
Dates: Start 2019-11-26 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of functional decline | 24 months
  assessed by short physical performance test battery
Incidence of injurious falls | 24 months
  assessed by fall questionnaire at each visit
Incidence of high blood pressure | 24 months
  Standardized blood pressure assessment in sitting position
Incidence of cognitive decline | 24 months
  assessed by Montreal Cognitive Assessment (MoCA)
Incidence of infections | 24 months
  assessed by infection questionnaire at each visit

SECONDARY OUTCOMES:
Incidence and prevalence of frailty | 24 months
  based on criteria by L. Fried (shrinking, weakness, poor endurance and energy, slowness, low physical activity level), SHARE-FI
Incidence and prevalence of impaired mobility | 24 months
  assessed by EQ5D-3L, physical activity questionnaire
Incidence and prevalence of functional dependency | 24 months
  assessed by PROMIS-HAQ
Incidence and prevalence of anemia or iron deficiency | 24 months
  assessed by blood markers (ferritin, soluble transferrin receptor, RBC, Hb, erythrocyte indices (MCV, MCH, MCHC), reticulocytes)
Incidence and prevalence of any cardiovascular disease | 24 months
  assessed by medical history
Incidence and prevalence of heart arrhythmia | 24 months
  assessed by ECG
Incidence and prevalence of atrial fibrillation | 24 months
  assessed by ECG
Incidence and prevalence of heart failure, cardiomyopathy, heart valves abnormalities | 24 months
  assessed by medical history, ECG, physical examination
Incidence of stroke | 24 months
  assessed by medical history
Incidence and prevalence of Type 2 diabetes | 24 months
  assessed by medical history
Incidence and prevalence of dementia | 24 months
  assessed by medical history
Incidence and prevalence of osteoarthritis | 24 months
  assessed by medical history
Incidence and prevalence osteoporosis | 24 months
  assessed by medical history
Incidence and prevalence of sarcopenia, osteosarcopenia | 24 months
  assessed by medical history
Incidence and prevalence of any gastrointestinal disease | 24 months
  assessed by medical history
Incidence and prevalence of gastroesophageal reflux disease (GERD) | 24 months
  assessed by medical history
Incidence and prevalence of any micronutrient deficiency (Vitamins, Minerals and fatty acids) | 24 months
  assessed by medical history
Incidence and prevalence of knee buckling | 24 months
  assessed by medical history, Buckling, KOOS, HOOS
Incidence and prevalence of chronic pain | 24 months
  assessed by medical history, McGill, Joint Map, EQ5D-3L
Incidence and prevalence of subjective memory complaints | 24 months
  assessed by medical history, MoCA, MACQ
Incidence and prevalence of hearing impairment | 24 months
  assessed by medical history, hearing test, physical examination
Incidence and prevalence of depression | 24 months
  assessed by medical history, GDS
Incidence and prevalence insomnia | 24 months
  assessed by medical history, Insomnia
Incidence and prevalence of chronic inflammation | 24 months
  assessed by medical history, blood marker (e.g. CRP)
Incidence and prevalence of polypharmacy | 24 months
  assessed by medication
Incidence and prevalence of inappropriate medication prescription | 24 months
  assessed by medication
Incidence and prevalence of age related morbidity by individual drug use (e.g. Proton-Pump-Inhibitors, anticoagulants, benzodiazepines, antibiotics) | 24 months
  assessed by medication
Incidence and prevalence of malnutrition | 24 months
  assessed by medical history, FFQ, GOHAI, Rome
Incidence and prevalence of urinary incontinence | 24 months
  assessed by medical history, IPPS, QUID
Incidence and prevalence of impaired quality of life | 24 months
  assessed by EQ5D-3L
Incidence and prevalence of functional decline | 24 months
  assessed by medical history
Incidence of fractures | 24 months
  assessed by fracture rate
Incidence of all-cause hospitalization | 24 months
  assessed by medical history
Incidence and prevalence of frequent health care utilization | 24 months
  assessed by medical history
trajectories of frequent health care utilization | 24 months
  assessed by medical history
Incidence of nursing home placement | 24 months
  assessed by medical history
Incidence of cancer (any cancer, gastro-intestinal, breast cancer in women, prostate cancer in men) | 24 months
  assessed by medical history
Incidence of all-cause mortality | 24 months
Prevalence of MIND diet adherence (DO-HEALTHcohort-MINDful substudy) | 24months
  assessed by FFQ
Prevalence and Incidence of Mild Cognitive impairment (DO-HEALTHcohort-MINDful substudy) | 24months
  assessed by MoCA
Dual-tasking gait variability (DO-HEALTHcohort-MINDful substudy) | one time
  assessed by GAITRite® Platinum (Basel only)
Prevalence of confirmed Covid-19 cases (DO-HEALTHcohort-MINDful substudy) | 24 months
  assessed by medical history
Prevalence of Covid-19 vaccinated participants (DO-HEALTHcohort-MINDful substudy) | 24 months
  assessed by medical history
Prevalence of reported subjective cognitive decline (DO-HEALTHcohort-MINDful substudy) | 24 months
  assessed by MAC-Q, GDS, EQ5D-3L
Covid-19 related resilience (DO-HEALTHcohort-MINDful substudy) | one time
  assessed by Brief Resilience Scale (BRS)
Covid-19 related stress (DO-HEALTHcohort-MINDful) | one time
  assessed by Covid-19 Pandemic Stress Scale (CPSS)
Covid-19 related coping behaviours (DO-HEALTHcohort-MINDful) | one time
  assessed by Pandemic Coping Scale (PCS)

CONTACTS AND LOCATIONS:
Overall Officials: Heike Bischoff-Ferrari, Prof. Dr. med. DrPH, Principal Investigator — University of Zurich
Locations (1):
- Centre on Aging and Mobility, University of Zurich, City Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No